CLINICAL TRIAL: NCT04383821
Title: Comparison of the Effects of Two Oxygen Delivery Systems on Arterial Blood Gases: Non-rebreather Mask Versus Double-trunk Mask
Brief Title: Comparison of the Non-rebreather Mask With the Double-trunk Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PT, PhD, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DTM-002
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-Trunk Mask (Experimental): The oxygen delivery system is the DTM
  Interventions: Device: Double-Trunk Mask
- Non-Rebreather Mask (Active Comparator): The oxygen delivery system is the NRM
  Interventions: Device: Non-Rebreather mask

INTERVENTIONS:
Device: Double-Trunk Mask — The DTM (oxygen delivery system) is worn by the patient for 30 minutes.
  Arms: Double-Trunk Mask
Device: Non-Rebreather mask — The NRM (standard oxygen delivery system) is worn by the patient for 30 minutes.
  Arms: Non-Rebreather Mask

SUMMARY:
This study will compare the impact of the Double-Trunk Mask (DTM) with the Non-Rebreather Mask (NRM) on the blood gases of patients with severe hypoxemia.

DETAILED DESCRIPTION:
The Double-Trunk Mask (DTM) is a device designed to increase the fraction of inspired oxygen in patients who receive oxygen therapy. The mask is composed of a regular aerosol mask with corrugated tubing (15 cm length) inserted into two lateral holes.

Each included patient will wear the standard Non-Rebreather Mask (NRM) which is the standard delivery oxygen system for patients with acute severe hypoxemia. Then the patients will wear the DTM for 30 minutes. Finally the DTM will be replaced by the NRM for the next 30 minutes. The impact of both oxygen delivery system will be assessed by measuring the change of blood gases with each system.

ELIGIBILITY:
Inclusion Criteria:

• Acute hypoxemia not corrected with nasal cannula

Exclusion Criteria:

* Chronic obstructive pulmonary disease or other chronic respiratory disease with hypercapnia
* Confusion
* Contra-indications to arterial blood gas sampling (peripheral arteriopathy, bleeding disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in PaO2 | At baseline and 30 minutes after wearing DTM
  Oxygen tension (PaO2) in mmHg will be analyzed from a sample taken from the arterial system

SECONDARY OUTCOMES:
Changes in PaCO2 | At baseline and 30 minutes after wearing DTM
  Carbon dioxide tension (PaCO2) in mmHg will be analyzed from a sample taken from the arterial system
Changes in pH | At baseline and 30 minutes after wearing DTM
  Potential of Hydrogen (pH) will be analyzed from a sample taken from the arterial system.
Changes in respiratory rate | At baseline and 30 minutes after wearing both systems
  Respiratory rate is measured during one minute by visual inspection.
Comfort with the oxygen delivery systems | 30 minutes after wearing both systems
  A Likert scale from -5 to +5 will be used to measure the subjective comfort of the patient while wearing both oxygen delivery systems
Dyspnea with the oxygen delivery systems | 30 minutes after wearing both systems
  A Visual Analogic Scale 0 to 10 will be used to measure the dyspnea of the patient while wearing both oxygen delivery systems

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels, Brussels Capital
  - Epicura, Hornu
  - Centre Hospitalier Universitaire de Tivoli, La Louvière